CLINICAL TRIAL: NCT05959889
Title: Evaluating the Effect of Montelukast on Doxorubicin Induced Cardiotoxicity in Breast Cancer Patients.
Brief Title: Effect of Montelukast on Doxorubicin Induced Cardiotoxicity in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Associate Professor, Damanhour University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Montelukast in Breast cancer
Record Dates: First submitted 2023-07-16; First posted 2023-07-25 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Doxorubicin Induced Cardiotoxicity
Keywords: Montelukast; Doxorubicin; Induced Cardiotoxicity; Breast cancer Patients
MeSH Terms: conditions — Breast Neoplasms | interventions — montelukast

STUDY DESIGN:
Intervention Model Description: a prospective, randomized (1:1) controlled trial that will be carried out on 50 patients who are candidate to evaluate the effect of montelukast on doxorubicin induced cardiotoxicity after 4 cycles of AC. Patients will be randomly allocated into two equal groups (25 patients each); group (A) for controlled (placebo), and group (B) for montelukast
Who Masked: Participant, Investigator
Masking Description: prospective, double blind randomized (1:1) controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): group (A) will recieved placebo tablet.
  Interventions: Other: Placebo
- Motelukast Group (Active Comparator): Patients will receive motelukast 10 mg for 4 cycles of AC.
  Interventions: Drug: Montelukast

INTERVENTIONS:
Other: Placebo — Patients will receive placebo tablets for 4 cycles of AC.
  Other Names: Placebo tablet
  Arms: Placebo Group
Drug: Montelukast — Patients will receive motelukast 10 mg for 4 cycles of AC.
  Other Names: Montelukast tablet
  Arms: Motelukast Group

SUMMARY:
This is a prospective, randomized (1:1) controlled trial that will be carried out on 50 patients who are candidate to evaluate the effect of montelukast on doxorubicin induced cardiotoxicity after 4 cycles of AC. Patients will be randomly allocated into two equal groups (25 patients each); group (A) for controlled (placebo), and group (B) for montelukast. Blood samples will be collected from the study subjects and analyzed for serum levels of the NF-KB and pro-BNP. Assessment of the biomarkers will be done at two time points: at baseline and after treatment with montelukast.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the effect of montelukast on doxorubicin induced cardiotoxicity in breast cancer patients through assessing serum NT-proBNP and NF-KB. The secondary objective is to evaluate the safety and side effects of montelukast on doxorubicin induced cardiotoxicity in breast cancer patients.

Methodology and study design:

1. Ethical committee approval will be obtained from Ethics committee of Faculty of Pharmacy, Damanhour University.
2. About 50 patients who are candidate to the study will be recruited from Damanhour Cancer Institute.
3. All participants will provide an informed consent.
4. Demographic data; age (year), sex (female/male), weight (kg), height (cm), BMI (kg/m2) will be collected.
5. About 5 ml of venous blood will be withdrawn by antecubital venipuncture from each participant at baseline and after receiving montelukast 10 mg once daily at bed time for 4 cycles of AC. At each time point blood samples will be collected into plain test tubes and centrifuged at 4500×g for 10 min and serum will be frozen at - 80 ◦C until analysis of the biomarkers using ELISA kits.
6. Montelukast tablets will be provided on monthly intervals and the participants' adherence will be assessed through the medications refilling rate. Participants will also be followed-up by weekly telephone calls and monthly direct meetings to assess their adherence and report any drug related adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age≥18 and≤ 70years old) with biopsy-confirmed diagnosis of breast cancer according to the American Joint Committee on Cancer (TNM staging system).
2. Patients with performance status (<2) according to Eastern Cooperative Oncology Group (ECOG).
3. Patients with adequate hematologic parameters (absolute neutrophil count≥1.5× 109/L, platelet count≥100× 109/L, hemoglobin level≥10 g/dl), adequate liver function (serum bilirubin<1.5 mg/dl), and adequate renal function (serum creatinine<1.5 mg/dl, creatinine clearance (CrCl)>45 ml/min).

Exclusion Criteria:

1. Patients who refuse to sign the written consent.
2. If blood cell counts are too low.
3. Severe liver problem.
4. Recent heart attack or have severe heart problems.
5. Previous treatment with Doxorubicin or certain other anticancer medications.
6. Allergy to certain other anti-cancer medicines, doxorubicin hydrochloride, Cis-platin, vincristine, paclitaxel, docetaxel, foscarnet, etc.

   in the last 6 months.
7. Women with evidence of metastasis at the initial assessment.
8. Presence of clinical evidence for severe cardiac illness (angina pectoris, uncontrolled hypertension, arrhythmias, and left ventricular ejection fraction<50%).
9. Pregnant and breast-feeding women.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
NF-KB | 6 months
  serum concentration of the NF-KB (ng/dl)
pro-BNP | 6 months
  serum concentration of the pro-BNP (ng/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Noha A. El bassiouny, Lecturer, Study Director — Damanhour University
Locations (1):
- Damanhour Oncology Center, Damanhūr, Elbehairah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Said MM, Bosland MC. The anti-inflammatory effect of montelukast, a cysteinyl leukotriene receptor-1 antagonist, against estradiol-induced nonbacterial inflammation in the rat prostate. Naunyn Schmiedebergs Arch Pharmacol. 2017 Feb;390(2):197-205. doi: 10.1007/s00210-016-1325-4. Epub 2016 Dec 1. PMID 27909742
- [Background] Elnoury HA, Elgendy SA, Baloza SH, Ghamry HI, Soliman M, Abdel-Aziz EA. Synergistic impacts of Montelukast and Klotho against doxorubicin-induced cardiac toxicity in Rats. Toxicol Res (Camb). 2022 Jun 20;11(4):592-604. doi: 10.1093/toxres/tfac023. eCollection 2022 Aug. PMID 36051669
- [Derived] Gomaa NF, Werida RH, El-Gowily AG, El-Bassiouny NA. Evaluating the role of montelukast on doxorubicin-induced cardiotoxicity in breast cancer patients. Support Care Cancer. 2025 Oct 1;33(10):897. doi: 10.1007/s00520-025-09947-z. PMID 41034674